CLINICAL TRIAL: NCT04641325
Title: Evaluating the Effects of Moderate Physical Activity on Health and Well-being in Adolescents and Young Adults With Marfan Syndrome
Brief Title: Marfan Syndrome Moderate Exercise Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Marfan Foundation (Other)
Responsible Party: Principal Investigator, Shaine Morris, Associate Professor, Pediatrics-Cardiology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-45475
Record Dates: First submitted 2020-04-23; First posted 2020-11-23 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Marfan Syndrome
Keywords: Cardiovascular; Moderate Exercise; Physical Therapy
MeSH Terms: conditions — Marfan Syndrome

STUDY DESIGN:
Intervention Model Description: The first part of trial was a Randomized Controlled Step-Wedge Pilot Trial as below 2 groups (Exercise Intervention Group and Current Care Group) The first phase of the study will maintain the Current Care Group as the control. At the end of the first phase, the Current Care Group will crossover and receive the Exercise Intervention as the second phase of the trial.
  With the COVID-19 pandemic causing delays in the study, and decreased enrollment and decreased access to MRI, the study was altered to a single group. comparing the same outcomes at baseline and after the intervention. This eliminates the blinding of the PI, but those interpreting the tests are still blinded.
Masking Description: The primary investigator and the co-PI (physical therapist) will know whether testing is at baseline or follow-up, but will not know the cardiovascular outcome measures. The cardiovascular outcomes assessor will be fully blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention Group (Experimental): Group of up to 20 patients will receive all of the preliminary outcome measure testing (cardiovascular, musculoskeletal, and psychological screening) in addition to exercise intervention education, demonstration, and follow up to ensure compliance and safety.
  Interventions: Other: Exercise Intervention Group

INTERVENTIONS:
Other: Exercise Intervention Group — Patients will be educated on methods of self-evaluating exertion and cardiovascular effort by assessing respiratory rate and perceived exertion. Next, patients will be given options for cardiovascular activities and complete at a moderate level of activity for a minimum of 150 minutes per week. Patients will perform a combination of exercises under the supervision of a physical therapist until a mod intensity level is reached and sustained. Patients will be taught to use the activity tracker to record their heart rate, activity, and PES. Patients will have a phone call every week to assess status, answer questions, and provide guidance on progressing intensity or duration of exercise. At the end of 8 weeks all patients will return for re-assessment.

SUMMARY:
Marfan syndrome (MFS) affects multiple organ systems including the heart, bones, ligaments, and eyes, and is associated with significant risk of aortic dissection. Given limited evidence from in-vitro studies, and theoretical concerns, the majority of patients with MFS are restricted from certain physical activities. The lack of exercise and deconditioning have detrimental effects including increasing weakness, joint pain, decreased endurance, and depressive symptoms. Given the significant paucity of data currently existing on the effects of exercise in humans with MFS, and the recent, optimistic findings in rodent models, this pilot trial was established to assess the effects of moderated dynamic exercise in adolescents and young adults with MFS.

DETAILED DESCRIPTION:
Marfan syndrome (MFS) affects multiple organ systems including the heart, bones, ligaments, and eyes, and is associated with significant risk of aortic dissection. Given anecdotal reports of aortic dissection, limited evidence from in-vitro studies, and theoretical concerns, the majority of patients with MFS are restricted from certain physical activities, most commonly isometric exercise and contact sports. Published guidelines also suggest restriction from highly dynamic competitive sports. While clinicians may mean to restrict patients only from competitive sports, often children and families interpret this caution as applying to almost all exercise, resulting in a large number of patients with Marfan syndrome being sedentary. This lack of exercise and deconditioning likely have detrimental effects in increasing weakness and joint pain and decreasing endurance. Depressive symptoms are also not uncommon in Marfan syndrome, and may be triggered or exacerbated by guidance to acutely cease participation in sports at the time of diagnosis.

To date, as far as the investigators are aware, there are no published controlled studies on the effects of dynamic exercise on human subjects. In 2017, Mas-Stachurska et al published a study suggesting that a moderate level of dynamic exercise mitigated progressive degradation of the cardiac structures typically seen in Marfan Syndrome in a rodent sample. This study suggests the possibility that the fears surrounding moderate exercise in humans may be unwarranted. In addition, this study suggests that moderate exercise may actually protect the aorta and myocardium, in addition to the numerous other physical and emotional benefits that have been shown to result from consistent exercise. The overall goal is to evaluate the effects of a moderate dynamic exercise program on measures of cardiovascular, muscular, and mental health in adolescents and young adults with Marfan syndrome. The investigators plan to perform a randomized pilot study to calculate effect estimates to perform a larger multi-center study. The objective is to 1) randomize 20 patients with Marfan syndrome age 12-21 years to current status (controls) versus a moderate dynamic exercise intervention, then 2) allow the control group patients to undergo the exercise intervention. The investigators will then compare outcomes between both the intervention and control groups, and between the baseline and post-intervention states. Specific outcome measures will include cardiovascular assessment: maximal oxygen uptake (max VO2), segmental and central aortic stiffness, ventricular mass and volume, and endothelial function, muscular/physical assessment: manual muscle testing (MMT), functional balance, and pain assessment, and quality of life/mental health assessment: health-related quality of life, depression and anxiety screening scales. The hypothesis is that the intervention of a moderate exercise program introduced by a licensed physical therapist will result in improvement in cardiovascular status, muscular health, and mental health without detrimental effects on the aortic wall.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 12-21
* Diagnosis of Marfan Syndrome
* Must not have other conditions that limit the patients ability to perform exercise

Exclusion Criteria:

* Patients who have undergone aortic surgery
* Patients with major congenital heart disease

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Maximum VO2 | 4 months
  Maximum VO2 in ml/kg/minute will be collected via Exercise Stress Test. Range 30-85, higher is better.

SECONDARY OUTCOMES:
Mean systolic blood pressure | 4 months
  mmHg, range 70-200, both low and high are abnormal, goal is age, sex and height-based, goal 10-50 percentile
Mean Diastolic blood pressure | 4 months
  mmHg, range 20-150, both low and high are abnormal, goal is age, sex and height-based, goal 10-50 percentile
Mean pulse pressure | 4 months
  mmHg, systolic blood pressure minus diastolic blood pressure, range 30-70 mmHg, goal is normal range for age and sex
Weight | 4 months
  kg, range 50-300kg, lower is better, excluding underweight patients
BMI | 4 months
  kg/m2, lower is better generally, excluding pts with BMI <5% for age
Left ventricular strain by cardiac MRI | 4 months
  Continuous measure derived from post-processing MRI
Right ventricular strain by cardiac MRI | 4 months
  Continuous measure derived from post-processing MRI
Aortic root strain | 4 months
  Continuous measure %, higher is less stiff, Range 0-40
Aortic Root Distensibility | 4 months
  ×10-3 mm Hg-1, Continuous measure, range 0.1-10
Aortic Root β-Stiffness index | 4 months
  No units, Range 0.1-90
Maximum aortic root dimension | 4 months
  Measured in cm, range 1-8cm
Aortic root z-score | 4 months
  No units, based on body surface area published references, range -3 to 25
Aortic pulse wave velocity from MRI | 4 months
  meters/second, range 0-30
Pulse wave velocity derived from applanation tonometry | 4 months
  meters/second, range 0-30
Augmentation index | 4 months
  %, range 1-90
Manual muscle testing score | 4 months
  Grade 0-5, higher is better
Reactive hyperemia index | 4 months
  no units, 0-4 range, higher is worse
Visual analog assessment of pain | 4 months
  no units, scale from 0-6, 6 is worse
Single Leg Stance Test | 4 months
  seconds, higher is better
Single limb squat test score | 4 months
  seconds, higher is better
Star Excursion Balance Test | 4 months
  %, range 0-100, higher is better
6M Timed Hop Test | 4 months
  milliseconds, range 1 to infinity, lower is better
Scale for Child Anxiety Related Emotional Disorders (SCARED) (ages 12-18 y) | 4 months
  41 item scale, each with 3 point Likert scale, scale is summed, range 0-123, higher is worse
Quality of Life Scale (QOLS) (ages 19-21 y) | 4 months
  16 items, each with 7 point Likert, higher is worse
Pediatric Quality of Life Scale (PedsQL) scale scores | 4 months
  reported in 3 domains, each reported on Likert scale, scaled to 0-100 scale, lower is worse
Children's Depression Inventory (CDI) 2 (ages 12-18 y) | 4 months
  28-item assessment that yields a Total Score, 2 scale scores, and 4 subscale scores. For each item, respondent is presented with 3 choices that correspond to 3 levels of symptomatology: 0 (absence of symptoms), 1 (mild or probable symptom), or 2 (definite symptom). Lower is better
Depression, Anxiety, & Stress Scale (DASS) (ages 19-21 y) | 4 months
  set of 3 self-report scales. Each scale contains 14 items, each with a 4-point severity/frequency scale, higher is worse

CONTACTS AND LOCATIONS:
Overall Officials: Shaine A Morris, MD MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No